CLINICAL TRIAL: NCT04604015
Title: RoBotic TCD Ultrasound BubbLe Study Compared to Transthoracic Echocardiography for Detection of Right to Left Shunt
Acronym: BUBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovaSignal Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NA-07BBL-01
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Embolic Stroke of Undetermined Source; Transient Ischemic Attack; Right-To-Left Atrial Shunt; Patent Foramen Ovale
MeSH Terms: conditions — Ischemic Attack, Transient; Foramen Ovale, Patent | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: The NeuralBot Investigational System is comprised of both the Lucid M1 System and the NeuralBot accessory. The NeuralBot accessory must be used with the Lucid M1 System and cannot operate independently. The NB-IS is a modification of a 510k cleared device called NeuralBot Guided Head mounted Accessory (K180455;22May2018). The NeuralBot Investigational System is the investigational study device used in this study.
  The NeuralBot Investigational System (NB-IS) moves two ultrasound probes around the two temporal regions (Right and Left) of the head to find the transtemporal window and then optimizes cerebral blood flow velocity (CBFV) measurements. The system uses TCD data to systematically specify and evaluate probe positions. The NeuralBot Investigational System consists of a head-support structure that houses two probe positioning modules, a robotic controller unit and computer tablets. The NeuralBot Investigational System is non-invasive and does not deliver energy into a subject.
Masking Description: All de-identified imaging data will be sent to a core laboratory which will provide independent quantitative and qualitative assessment of all NB-IS TCD and Standard of care (SOC) TCD, TTE, and TEE bubble study data. They will be blinded to the study and local diagnostic report data and provide independent review. The Core Lab interpretations will supersede all local interpretations and will be applied to all study endpoint analyses as applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- NeuralBot Investigational System/TTE Std of Care (Experimental): Investigational Robotic Transcranial Doppler (TCD)/TTE Std of Care
  Interventions: Diagnostic Test: NeuralBot Investigational System; Diagnostic Test: Transthoracic Echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: NeuralBot Investigational System — The NeuralBot Investigational System when used with the Lucid M1 System is a medical ultrasound device which assists the user in the setup and acquisition of cerebral blood flow velocity via the patient's temporal windows. It is intended for use as an adjunct to standard clinical practices for measuring and displaying cerebral blood flow velocity and the occurrence of transient emboli within the blood stream.
  Other Names: Lucid Robotic System; NovaGuide; Lucid TCD; NovaBot
Diagnostic Test: Transthoracic Echocardiography (TTE) — A test that uses ultrasound to create a hemodynamic assessment for major cardiovascular events.
  Other Names: TTE

SUMMARY:
This study is a multi-center, prospective, single-arm, non-significant risk (NSR) device study in which up to 150 evaluable subjects with suspicion of embolic stroke of undetermined source (ESUS) will be evaluated with NB-IS TCD and standard of care TTE to screen for right to left shunt (RLS) or patent foramen ovale (PFO). Additionally, up to 150 evaluable subjects will be evaluated with NB-IS TCD and standard of care TEE.

DETAILED DESCRIPTION:
The objectives of the study is to evaluate the shunt detection rate of the NeuralBot Investigational System (NB-IS) TCD relative to standard of care diagnostic techniques (transthoracic echocardiography (TTE), transesophageal echocardiography (TEE), and standard transcranial Doppler ultrasound (TCD) and to assess the safety, accuracy and usability of the NB-IS device.

ELIGIBILITY:
Inclusion Criteria TTE Main Study:

1. Subject 18 years of age and older.
2. Subject presents with a clinical condition characterized by neurological signs and symptoms that, in the opinion of the investigator, include embolic stroke or transient ischemic attack (TIA) in the differential diagnosis.
3. Scheduled for a transthoracic echocardiograph (TTE) study with agitated saline contrast (bubble study) per standard of care within ±30 days of informed consent.
4. Subject is able to successfully perform a Valsalva Maneuver (VM).
5. Subject or Legally Authorized Representative has the ability to provide informed consent and comply with the protocol.

Exclusion Criteria TTE Main Study:

1. Subject has undergone a right to left shunt (RLS) or patent foramen ovale (PFO) closure.
2. Female who is pregnant or lactating at time of admission
3. Subjects who underwent partial or full craniotomy/craniectomy within the past 6 months.
4. Subjects who have a physical limitation preventing TCD headset placement

Inclusion Criteria TEE Sub-Study (after first 150 subjects in Main TTE study enrolled):

1. Subject 18 years of age and older.
2. Subject presents with a clinical condition characterized by neurological signs and symptoms that, in the opinion of the investigator, include embolic stroke or TIA in the differential diagnosis.
3. Scheduled for a transesophageal echocardiograph (TEE) study with agitated saline contrast (bubble study) per standard of care within ±30 days of informed consent.
4. Subject is able to successfully perform a Valsalva Maneuver (VM).
5. Subject or Legally Authorized Representative has the ability to provide informed consent and comply with the protocol.

Exclusion Criteria TEE Sub-Study (after first 150 subjects in Main TTE study enrolled):

1. Subject has undergone a right to left shunt (RLS) or patent foramen ovale (PFO) closure.
2. Female who is pregnant or lactating at time of admission
3. Subjects who underwent partial or full craniotomy/craniectomy within the past 6 months.
4. Subjects who have a physical limitation preventing TCD headset placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Alexandrov, MD, Study Chair — The University of Tennessee Health Science Center; Mark Rubin, MD, Principal Investigator — The University of Tennessee Health Science Center
Locations (7):
- United States (7):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Providence Brain & Spine Institute, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - CHI Memorial Hospital, Chattanooga, Tennessee
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - Houston Methodist Neurological Institute, Houston, Texas
  - Swedish Hospital, Seattle, Washington

REFERENCES:
- [Result] Rubin MN, Shah R, Devlin T, Youn TS, Waters MF, Volpi JJ, Stayman A, Douville CM, Lowenkopf T, Tsivgoulis G, Alexandrov AV. Robot-Assisted Transcranial Doppler Versus Transthoracic Echocardiography for Right to Left Shunt Detection. Stroke. 2023 Nov;54(11):2842-2850. doi: 10.1161/STROKEAHA.123.043380. Epub 2023 Oct 5. PMID 37795589
- See also: Robot-Assisted Transcranial Doppler Versus Transthoracic Echocardiography for Right to Left Shunt Detection — https://pubmed.ncbi.nlm.nih.gov/?term=Robot+assisted+Transcranial+Doppler+versus+transthoracic

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 154 subjects were enrolled (signed Informed Consent), 129 evaluable and 121 completed the protocol.
Groups:
- NeuralBot Investigational System/TTE Std of Care: Subjects presented with suspected embolic cerebrovascular event, were scanned by both devices within 30 days of the index scan.
Period: Overall Study
Arm/Group | NeuralBot Investigational System/TTE Std of Care
Started | 154
Completed | 121
Not Completed | 33
Not completed — Incomplete Data Collection | 33

BASELINE CHARACTERISTICS:
Population: Per Protocol/Completed subjects
Groups:
- NeuralBot Investigational System: Robotic TCD monitoring during bubble exam
  NeuralBot Investigational System: The NeuralBot Investigational System when used with the Lucid M1 System is a medical ultrasound device which assists the user in the setup and acquisition of cerebral blood flow velocity via the patient's temporal windows. It is intended for use as an adjunct to standard clinical practices for measuring and displaying cerebral blood flow velocity and the occurrence of transient emboli within the blood stream.
Arm/Group | NeuralBot Investigational System
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 103
  More than one race | 0
  Unknown or Not Reported | 4
Stroke diagnosis [Count of Participants; unit: Participants]
  Embolic stroke undetermined source | 68
  Transient ischemic attack | 9
  Other (not specificed) | 44
  Absent transtemporal windows | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Detection of Right to Left Shunt (RLS)/Patent Foramen Ovale (PFO) Using Robotic Assisted TCD (Study Device)
Description: The primary outcome measure was the percent detection of Right to Left Shunt using the robotic assisted TCD (study device) and compare it to the percent detection of Right to Left Shunt using standard of care Transthoracic Echocardiography (TTE) for the same patient cohort. The detection of the Right to Left Shunt included site and independent Core Lab assessment of TTE.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | NeuralBot Investigational System/TTE Std of Care
Number analyzed (Participants) | 121
Participants
  NeuralBot Investigational System: Positive | 74
  NeuralBot Investigational System: Negative | 47
  TTE standard of care: Positive | 24
  TTE standard of care: Negative | 97
Statistical Analysis 1: Comparison: NeuralBot Investigational System/TTE Std of Care; The study was powered based on the results of a meta-analysis reporting the pooled NeuralBot (TCD) sensitivity for Right to Left Shunt detection, and the pooled TTE sensitivity for Right to Left Shunt detection; Test type: Other; p < 0.001, McNemar; absolute difference = 41, 95% CI 2-sided [32.9 to 50.2]

ADVERSE EVENTS:
Time Frame: Device related adverse events were collected during the period of device use (1 Day)
Description: Device related events (only) were collected during the period of device use.
Groups:
- NeuralBot Investigational System: Investigational Robotic Transcranial Doppler (TCD)
  NeuralBot Investigational System: The NeuralBot Investigational System when used with the Lucid M1 System is a medical ultrasound device which assists the user in the setup and acquisition of cerebral blood flow velocity via the patient's temporal windows. It is intended for use as an adjunct to standard clinical practices for measuring and displaying cerebral blood flow velocity and the occurrence of transient emboli within the blood stream.
- TTE Std of Care: Control Device- Transthoracic Echocardiography
  Transthoracic Echocardiography (TTE): A test that uses ultrasound to create a hemodynamic assessment for major cardiovascular events.
Arm/Group | NeuralBot Investigational System | TTE Std of Care
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/121
Other Adverse Events (participants affected / at risk) | 0/121 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT04604015/Prot_SAP_000.pdf